CLINICAL TRIAL: NCT01248130
Title: Omega-3 Fatty Acids Monotherapy in Children and Adolescents With Autism Spectrum Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a change in the research priorities of the principal investigator in combination with low subject interest.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Clinical Investigator, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-P-001593
Record Dates: First submitted 2010-11-19; First posted 2010-11-25 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Omega-3 Fatty Acid; Autism Spectrum Disorders; Pervasive Developmental Disorders; Children; Cognitive Functioning
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Fatty Acid Treatment (Active Comparator)
  Interventions: Drug: Omega-3 Fatty Acid
- Placebo (Sugar Pill) (Placebo Comparator)
  Interventions: Drug: Omega-3 Fatty Acid

INTERVENTIONS:
Drug: Omega-3 Fatty Acid — Children with Autism Spectrum Disorders will be randomized to receive either 1500mg (3 capsules) omega-3 fatty acids or placebo. Each 500mg capsule contains 350mg EPA and 50mg DHA. Omega-3 fatty acids dosing will be on a forced titration schedule to 3 capsules per day. All subjects will start with 1 capsule per day with an increase to 3 capsules per day by week 2. Subjects will be maintained at 3 capsules per day thereafter until the end of the trial (completion/discontinuation). During the 12 weeks of the study period, participants will be evaluated at weekly intervals during the first three weeks of the trial (baseline, weeks 1-3) and tri-weekly thereafter till the end of the trial (weeks 6, 9 and 12). At each visit, measures of safety and effectiveness will be administered and subjects will be evaluated for response and side effects to the treatment. Study medications will be prescribed under double blind conditions.
  Other Names: Fish Oil

SUMMARY:
The primary aim of this study is to examine the efficacy and tolerability of short-term omega-3 fatty acids monotherapy in youth with Autism Spectrum Disorders (ASD). The investigators hypothesize that Omega-3 fatty acids will be efficacious in improving the core and associated features of ASD in youth, and that Omega-3 fatty acids monotherapy will be safe and well tolerated by youth with ASD. The secondary aim of this study is to examine the neuropsychological effect of Omega-3 fatty acids monotherapy in youth with ASD. The investigators hypothesize that omega-3 fatty acids will be efficacious in improving cognitive functions in youth with ASD.

ELIGIBILITY:
Inclusion

1. Male or female participants between 6 and 17 years of age, inclusive.
2. Fulfills diagnosis of autism spectrum disorders by meeting DSM-IV-TR PDD diagnostic criteria of autistic disorder, Asperger's disorder, or PDD-NOS as established by clinical interview assisted by MGH PDD Symptom Checklist.
3. Participants with at least moderate symptom severity of ASD as reflected by SRS score ≥ 85 and CGI-PDD severity score of ≥ 4 (moderately ill).
4. Subjects must be psychotropic drug-free for a minimum of four weeks prior to the baseline visit.
5. Subjects with mood, anxiety, or disruptive behavior disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.

Exclusion

1. I.Q. < 85.
2. DSM-IV-TR PDD diagnoses of Rett's disorder, and childhood disintegrative disorder.
3. Current diagnosis of a psychotic disorder or unstable mood or anxiety disorders as determined by the clinician.
4. Subject with marked severity of symptoms as suggested by the score of ≥ 5 (markedly ill) on CGI severity subscale for respective comorbid psychiatric disorders.
5. Clinically unstable psychiatric condition judged to be at a serious risk to self or others as determined by the clinician.
6. History of substance use (except nicotine or caffeine) within past 3 months, determined to be clinically significant by clinician.
7. Urine drug screen positive for substances of abuse.
8. Non-febrile seizures without a clear and resolved etiology in last month.
9. Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including:

   1. Pregnant or nursing females;
   2. Organic brain disorders;
   3. Uncorrected hypothyroidism or hyperthyroidism, as determined by study clinician;
   4. Untreated and/or unstable diabetes;
   5. Subjects with a clinically significant abnormality according to cardiology consultation (ECGs with clinically concerning intervals including PR, QTC, QRS, will be reviewed by cardiology).
   6. History of renal or hepatic impairment determined to be clinically significant by clinician.
10. Serious, unstable systemic illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease, as determined by clinician.
11. Any other concomitant medication with primary central nervous system activity other than specified in the Concomitant Medication section of the protocol.
12. Subjects who have difficulty swallowing pills.
13. History of known allergy to Omega-3 fatty acids, multiple drug allergies, or severe allergies.
14. A non-responder of, or history of intolerance to Omega-3 fatty acids, after treatment at an adequate dose and duration as determined by the clinician.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega-3 Fatty Acid Treatment | Placebo (Sugar Pill)
Started | 3 | 4
Completed | 1 | 4
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acid Treatment | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Social Responsiveness Scale (SRS) Total Raw Score
Description: The SRS is a 65-item rating scale completed by the participants parent or guardian. The scale measures the severity of autism spectrum symptoms as the occur in natural social settings. The total raw score is calculated by summing the 65 items. Total scores range from 0 to 195, where higher scores indicate greater severity. The outcome reported reflects the change from baseline (pre-treatment) in SRS Total raw score. When examining change from baseline, negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Pre-treatment - 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 Fatty Acid Treatment | Placebo (Sugar Pill)
Number analyzed (Participants) | 1 | 4
score on a scale | 0 (NA) — Only 1 participant in this Arm. | -7 (15.0)

2. Secondary Outcome: Change in NIMH Clinical Global Impression Scale for Pervasive Developmental Disorders (CGI-PDD) Improvement Scores
Description: The CGI-PDD Improvement scale is a clinician-rated assessment of the participant's improvement in symptoms compared to baseline. The CGI-PDD-I is rated on a scale of one (very much improved) to seven (very much worse) and values of zero (not assessed) are assigned to all participants at baseline. The outcome reported reflects the change in improvement score from baseline, where lower scores indicate greater improvement compared to baseline.
Time Frame: Pre-treatment - 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 Fatty Acid Treatment | Placebo (Sugar Pill)
Number analyzed (Participants) | 1 | 4
score on a scale | 4 (NA) — Only 1 participant in this Arm. | 3.3 (1.0)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Spontaneously reported AEs
Arm/Group | Omega-3 Fatty Acid Treatment | Placebo (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acid Treatment (N=3) | Placebo (Sugar Pill) (N=4)
Tiredness (General disorders) | 1 (1) | 0 (0)
Allergic reaction in eye (Immune system disorders) | 1 (1) | 0 (0)
Decreased energy (General disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
More isolative (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cold (Immune system disorders) | 0 (0) | 1 (2)
Broke left wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to a change in the research priorities of the Principal Investigator in combination with low subject interest. Therefore, no data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes